CLINICAL TRIAL: NCT05295199
Title: The Effect of Progressive Relaxation Exercise on Fatigue and Comfort Level After Major Orthopedic Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Aksaray University (Other)
Responsible Party: Principal Investigator, Funda Cetinkaya, Principal Investigator, Aksaray University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2020/01-24
Record Dates: First submitted 2022-03-10; First posted 2022-03-25 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Orthopedic Surgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Routine maintenance and Progressive relaxation exercise
  Interventions: Other: Progressive relaxation exercise
- Control (No Intervention): Routine maintenance

INTERVENTIONS:
Other: Progressive relaxation exercise — Progressive relaxation exercise is a type of exercise that involves voluntary stretching and relaxation of major muscle groups in the human body, from the hands to the feet.
  Arms: Experimental

SUMMARY:
This study was planned to determine the effect of progressive relaxation exercise to be applied after major orthopedic surgery on post-operative fatigue and comfort level.

DETAILED DESCRIPTION:
The symptom of fatigue causes tension, anxiety, fear, and insomnia in the person. Fatigue also negatively affects the comfort level of the patient along with the symptoms experienced in individuals.Suggestions and evaluations of the professional healthcare team, especially nurses, are of great importance in the effective fight against fatigue of patients.In this study, it is carried out to determine the effect of progressive relaxation exercise applied after major orthopedic surgery on fatigue and comfort level.

Hypothesis

H1: Progressive relaxation exercise to be applied after major orthopedic surgery reduces the post-operative fatigue level of patients.

H2: Progressive relaxation exercise to be applied after major orthopedic surgery positively affects the comfort level of the patients.

ELIGIBILITY:
Inclusion Criteria:

* The patients included in the study have undergone major orthopedic surgery (total knee or hip replacement, atroscopic surgery, vertebral surgery, shoulder surgery, amputation, etc.), Patients aged 18 and over Absence of speech and hearing problems Speak and understand Turkish

Exclusion Criteria:

* Being diagnosed with a psychiatric disorder, A complication developed in the patients before, during and three days after the operation,

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-03-10 (Actual); Primary Completion 2022-08-30 (Estimated); Study Completion 2022-08-30 (Estimated)

PRIMARY OUTCOMES:
General Comfort Scale | 1st day after surgery
  It is a scale developed to determine the comfort levels of patients.The lowest possible score is 48, the median score is 120, and the highest score is 192. As the score obtained from the scale increases, the level of comfort perceived by the patient increases.
Postoperative Fatigue Scale | 1st day after surgery
  It is a scale created to evaluate the post-operative fatigue level of patients.

SECONDARY OUTCOMES:
General Comfort Scale | 4th day after surgery
  It is a scale developed to determine the comfort levels of patients.The lowest possible score is 48, the median score is 120, and the highest score is 192. As the score obtained from the scale increases, the level of comfort perceived by the patient increases.
Postoperative Fatigue Scale | 4th day after surgery
  It is a scale created to evaluate the post-operative fatigue level of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Funda CETINKAYA, Principal Investigator — Aksaray University
Locations (1):
- Aksaray University, Aksaray, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No